CLINICAL TRIAL: NCT01120743
Title: Correlation Between Release of Cytokines From Liver Graft and Hemodynamic Stability During Liver Transplantation
Brief Title: Correlation Between Release of Cytokines From Liver Graft and Hemodynamic Instability
Status: Completed | Type: Observational
Sponsor: Penn State University (Other)
Responsible Party: Sponsor
Other Study IDs: No 28764
Record Dates: First submitted 2010-05-03; First posted 2010-05-11 (Estimated); Last update posted 2017-11-24 (Actual); Status verified 2017-11

CONDITIONS: Liver Transplantation
Keywords: liver failure; cytokines; hemodynamic instability
MeSH Terms: conditions — Liver Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood samples were obtained. All blood samples were placed on ice and processed with centrifugation. The plasma supernatant was frozen at -80º Celsius.
Oversight: Data Monitoring Committee: No

SUMMARY:
The primary goal of this project is to identify the source of cytokines that are released into circulation during graft reperfusion. Seventeen patients scheduled to have adult cadaveric liver transplantation at the Milton S. Hershey Medical Center were contacted as prospective participants. Blood samples were obtained from the radial artery, the portal vein, and from the graft irrigation. The level of pro-inflammatory cytokines was verified and compared with the amount of catecholamines used to maintain hemodynamic stability.

DETAILED DESCRIPTION:
Reperfusion of the graft is the most critical part of liver transplantation because of the difficulties in managing the resulting severe hemodynamic instability. The patients who are accepted to be listed for liver transplantation undergo evaluation of their cardiac function and are usually relatively stable with, at most, minimal cardiac problems (a requirement for inclusion in the liver transplantation program). Additionally, we observe completely unpredictable hemodynamic reactions during and after the graft reperfusion, requiring vastly different doses of catecholamine in order to maintain an acceptable level of perfusion pressure. The adverse cardiopulmonary effects are thought to be associated with the preexisting level of various proinflammatory factors, including cytokines (TNF-alpha, IL-6) and proinflammatory phospholipase A2 (sPLA2) produced in the graft as a reaction to the conservation solution and cold temperature (necessary to keep the organ capable for transplantation) and released into the bloodstream during reperfusion. The massive release of cytokines after unclamping of the graft may be responsible for negative inotropy and significant vasodilatation.

ELIGIBILITY:
Inclusion Criteria:

* All adult patients scheduled for liver transplantation will be offered the opportunity to participate in this research.

Exclusion Criteria:

* Patients unable or unwilling to provide adequate informed consent will be excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Study will include adult patients with end-stage liver disease accepted for liver transplantation.
Sampling Method: Non-Probability Sample
Enrollment: 17 (Actual)
Dates: Start 2008-08; Primary Completion 2010-04 (Actual); Study Completion 2010-04 (Actual)

PRIMARY OUTCOMES:
Measurement of cytokine levels (TNF-alpha, IL-1, Il-2, IL-6, IL-8) in the portal vein, radial artery and "flush" (from irrigation of the liver used to remove preservation solution from the liver graft) blood. | A period of 20 minutes, beginning at the start of reperfusion and continuing until 20 minutes after reperfusion.
  Cytokines released from the liver graft could be a cause for negative inotropy and systemic vasodilatation.

SECONDARY OUTCOMES:
Correlation between the level of cytokines and hemodynamic stability during reperfusion. | A period of 20 minutes, beginning at the start of reperfusion and continuing until 20 minutes after reperfusion.
  First 20 minutes after liver graft reperfusion is a time of maximal hemodynamic instability. A correlation between the level of cytokines and hemodynamic instability could be important for understanding of this condition

CONTACTS AND LOCATIONS:
Overall Officials: Dmitri Bezinover, MD, PhD, Principal Investigator — Penn State Milton S. Hershey Medical Center, Penn State College of Medicine
Locations (1):
- Penn State Milton S. Hershey Medical Center, Penn State College of Medicine, Hershey, Pennsylvania, United States

REFERENCES:
- [Derived] Bezinover D, Kadry Z, McCullough P, McQuillan PM, Uemura T, Welker K, Mastro AM, Janicki PK. Release of cytokines and hemodynamic instability during the reperfusion of a liver graft. Liver Transpl. 2011 Mar;17(3):324-30. doi: 10.1002/lt.22227. PMID 21384515